CLINICAL TRIAL: NCT05202158
Title: A Novel Method for Stone Area Sterilization During Retrograde Intrarenal Surgery (RIRS)
Brief Title: A Novel Method for Retrograde Intrarenal Surgery (RIRS)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ankara Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Ali Kaan Yildiz, Principal Investigator, Ankara Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RIRS2022
Record Dates: First submitted 2022-01-10; First posted 2022-01-21 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Kidney Stone
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Irrigation + Genta (Active Comparator): Patients treated with gentamicin in irrigation fluid during RIRS
  Interventions: Procedure: Addition of gentamicin to irrigation fluid during RIRS
- Irrigation (Sham Comparator): Patients treated only irrigation fluid during RIRS
  Interventions: Procedure: Only irrigation fluid during RIRS

INTERVENTIONS:
Procedure: Addition of gentamicin to irrigation fluid during RIRS — During the RIRS, the access sheath is placed first for security. Then, the stone in the kidney is detected with flexible URS and fragmented with a holmium laser. In this group of patients, 80 mg of gentamicin will be added to 3 liters of irrigation fluid while the stone is being fragmented.
  Arms: Irrigation + Genta
Procedure: Only irrigation fluid during RIRS — During the RIRS, the access sheath is placed first for security. Then, the stone in the kidney is detected with flexible URS and fragmented with a holmium laser. In this group of patients, only irrigation fluid will be used while the stone is fragmented.
  Arms: Irrigation

SUMMARY:
In this prospective randomised controlled study, investigators aims to evaluate the effect of 80 mg gentamicin added to 3 liters of irrigation fluid on stone free rate, intraoperative and postoperative complications during RIRS for kidney stones.

DETAILED DESCRIPTION:
Current advances in endoscopic technology for the upper urinary tract have expanded the diagnosis and treatment options for kidney stones. Retrograde intrarenal surgery (RIRS), defined as the use of effective lithotripters such as flexible ureteroscopes (fURSs) and holmium:yttrium aluminum garnet (holmium:YAG) lasers for intrarenal pelvic diseases, is a safe and effective, versatile and minimally invasive procedure for the kidney. . Current guidelines for the treatment of kidney stones recommend RIRS first for stones <2 cm. and RIRS as one of the first two options for stones >2 cm.. In studies dealing with kidney stones larger than 2 cm, the RIRS showed a cumulative stone-free success of 91%, but a complication rate of 8.6%. Of these, 44% were found to be ≥ Clavien 3 complications. In kidney stone endourological treatments, stone culture was found to be more effective in predicting complications than midstream urine culture. Even if the preoperative midstream urine culture is sterile, complication rates increase if there is bacterial growth in the stone culture in kidney stone surgery. Therefore, although complication rates are generally low, several concerns have arisen. In our study, the investigators aims to evaluate the effect of 80 mg gentamicin added to 3 liters of irrigation fluid on stone free rate and complications during RIRS for kidney stones.

ELIGIBILITY:
Inclusion Criteria:

* <2 cm. kidney stones

Exclusion Criteria:

* Ureteral stricture
* Active urinary tract infection
* Coagulopathies

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2022-02-15 (Actual); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Rate of postoperative complications | One year
  Rate of patients who had an complication after the operation

CONTACTS AND LOCATIONS:
Overall Officials: Ali Kaan Yildiz, Principal Investigator — Ankara Training and Resarch Hospital
Locations (1):
- Ankara Training and Research Hospital, Ankara, Altindag, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Turk C, Petrik A, Sarica K, Seitz C, Skolarikos A, Straub M, Knoll T. EAU Guidelines on Diagnosis and Conservative Management of Urolithiasis. Eur Urol. 2016 Mar;69(3):468-74. doi: 10.1016/j.eururo.2015.07.040. Epub 2015 Aug 28. PMID 26318710
- [Result] Walton-Diaz A, Vinay JI, Barahona J, Daels P, Gonzalez M, Hidalgo JP, Palma C, Diaz P, Domenech A, Valenzuela R, Marchant F. Concordance of renal stone culture: PMUC, RPUC, RSC and post-PCNL sepsis-a non-randomized prospective observation cohort study. Int Urol Nephrol. 2017 Jan;49(1):31-35. doi: 10.1007/s11255-016-1457-y. Epub 2016 Nov 15. PMID 27848063